CLINICAL TRIAL: NCT06662292
Title: Using Existing Social Ties to Promote Physical Activity: Effects of Digitally Delivered Team Social Support Training
Brief Title: Mobile Supportive Teams for Reinforcing Increased Daily Exercise Study
Acronym: STRIDES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Courtney Monroe, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00133610; R01DK138115 (NIH)
Record Dates: First submitted 2024-10-22; First posted 2024-10-28 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Physical Activity
Keywords: physical activity; exercise; adults; social support; smartphone; electronic health; mobile health; teams
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Team Program (Active Comparator): Teams randomized to this arm will be provided with personal physical activity goals focused on moderate-to-vigorous intensity aerobic physical activity minutes and steps. They will also be provided with a Fitibt wearable smartwatch for self-monitoring physical activity, receive weekly electronic feedback for the first month of the intervention about their physical activity progress, and have access to a mobile-compatible study web app containing behavior change content and physical activity progress information.
  Interventions: Behavioral: Mobile STRIDES app (psychoeducation features); Behavioral: Mobile STRIDES app (self-regulation features)
- Team+Training Program (Experimental): Teams randomized to this arm will receive the same intervention as the Team study arm, as well as digitally delivered social support training.
  Interventions: Behavioral: Mobile STRIDES app (psychoeducation features); Behavioral: Mobile STRIDES app (self-regulation features); Behavioral: Mobile STRIDES app (social support training features)

INTERVENTIONS:
Behavioral: Mobile STRIDES app (psychoeducation features) — Twelve theory-based physical activity behavior change lessons/modules during the course of the 3-month intervention.
Behavioral: Mobile STRIDES app (self-regulation features) — Personalized physical activity goals focused on moderate-to-vigorous intensity aerobic physical activity and steps. Physical activity (tracked with a Fitbit wearable smartwatch and synced with the Mobile STRIDES app) tracking component, displaying team and individual progress. Weekly individualized feedback messages crafted by a trained professional for the first month of the intervention.
Behavioral: Mobile STRIDES app (social support training features) — For the experimental group, the Mobile STRIDES app also includes five social support training lessons/modules (during the course of the 3-month intervention) focused on providing guidance related to effective communication when exchanging social support for physical activity within a team. In addition, six team feedback messages will be delivered to respective teams throughout the course of the 3-month intervention to reinforce content taught via the training lessons/modules. A weekly poll will also be administered that complements the social support training lessons, with cumulative results displayed.
  Arms: Team+Training Program

SUMMARY:
The goal of this research is to examine the addition of a digitally delivered social support training approach to an existing digital program designed to promote a physically active lifestyle among self-selected teams of adults who are not meeting physical activity guidelines. The main aims are to:

1. Determine if the social support training intervention promotes significantly greater changes in moderate-to-vigorous intensity aerobic physical activity (such as a brisk walk) as measured by an accelerometer (research grade physical activity measurement device) at 3 months compared to the same intervention without social support training among self-selected teams of adults who are not meeting the physical activity guidelines.
2. Determine if the social support training intervention promotes significantly greater changes in social support, motivation, accountability, and autonomy social support (free from excessive control and encouraging one's free will) at 3 months and 12 months compared to the same intervention without social support training.
3. Determine if the social support training intervention promotes significantly greater changes in moderate-to-vigorous intensity aerobic physical activity as measured by an accelerometer at 12 months compared to the same intervention without social support training.
4. Explore whether social support mediates increased and sustained moderate-to-vigorous intensity aerobic physical activity among the entire sample of participants.

DETAILED DESCRIPTION:
Self-selected teams of 3-8 insufficiently active adults (about 60 teams comprised of a total of 300 participants) will be randomized to receive either a 3-month, theory-based, technology-delivered physical activity intervention characterized by personalized physical activity goals, a wearable physical activity tracker, electronic feedback, and behavior change modules embedded within a mobile-compatible app (Team) or the same intervention plus digitally delivered social support training (Team+Training). Outcome assessments will be completed at baseline, 3, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

* be at least 18 years of age
* be insufficiently physically active (< 150 minutes per week of moderate-intensity equivalent aerobic physical activity as measured by waist-worn accelerometer (research grade physical activity measurement device) - i.e., sum of time spent in minutes of moderate-intensity activity plus twice the minutes spent in vigorous-intensity activity < 150 minutes per week)
* be part of a self-selected team of 3-8 individuals each of whom also meet all other eligibility criteria (members of the same household are only eligible to participate if they are on the same team - limit one team per household)
* have access to a smartphone (Android or iphone operating system-based) with an internet connection
* report being able to walk at least ¼ mile without stopping
* be able to provide informed consent
* complete all screening and baseline questionnaires and activities

Exclusion Criteria:

* participating in another physical activity study or program
* are pregnant, breastfeeding, less than 6 months post-partum, or plan to become pregnant during the time frame of the investigation
* report a medical condition that would affect the safety and/or efficacy of a physical activity program (e.g., terminal illness; uncontrolled heart condition, dementia, bulimia nervosa or binge eating disorder, other significant psychiatric problems, or use of insulin)
* report conditions that in the judgment of the Principal Investigator would render them unlikely to be able to independently follow the intervention protocol for 3 months, including conditions which might compromise their ability to engage independently with the intervention website materials and wearable physical activity tracker, as well as complete online questionnaires and adhere to wearing an accelerometer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in minutes per week of moderate-to-vigorous intensity aerobic physical activity (MVPA) at 3 months | Baseline and 3 months
  Change in minutes per week of moderate-to-vigorous intensity aerobic physical activity (MVPA) from baseline to 3 months as measured by accelerometer

SECONDARY OUTCOMES:
Change in minutes per week of moderate-to-vigorous intensity aerobic physical activity (MVPA) at 12 months | 3 months and 12 months
  Change in minutes per week of moderate-to-vigorous intensity aerobic physical activity (MVPA) from 3 months to 12 months as measured by accelerometer
Change in supportive accountability at 3 months | Baseline and 3 months
  Support Accountability Inventory adapted for physical activity and to query about one's team. Items rated on a Likert scale response format ranging from 1 (Strongly Disagree) to 7 (Strongly Agree) with a not applicable option, with higher total scores indicating higher perceived supportive accountability.
Change in motivation at 3 months | Baseline and 3 months
  Treatment Self-Regulation Questionnaire adapted for physical activity. Items scored using a 7-point Likert scale (1 = not at all to 7 = very true). Higher scores on the Autonomous Subscale indicate greater autonomous motivations for behavior change and higher scores on the Controlled Motivations subscale indicate higher controlled regulation.
Change in supportive accountability at 12 months | 3 months and 12 months
  Support Accountability Inventory adapted for physical activity and to query about one's team. Items rated on a Likert scale response format ranging from 1 (Strongly Disagree) to 7 (Strongly Agree) with a not applicable option, with higher total scores indicating higher perceived supportive accountability.
Change in motivation at 12 months | 3 months and 12 months
  Treatment Self-Regulation Questionnaire adapted for physical activity. Items scored using a 7-point Likert scale (1 = not at all to 7 = very true). Higher scores on the Autonomous Subscale indicate greater autonomous motivations for behavior change and higher scores on the Controlled Motivations subscale indicate higher controlled regulation.
Change in autonomy support at 3 months | Baseline and 3 months
  Important Other Climate Questionnaire adapted for physical activity and to query about one's team. Items rated on a Likert scale response format ranging from 1 (Strongly Disagree) to 7 (Strongly Agree) with a not applicable option, with higher total scores indicating higher perceived autonomy support.
Change in autonomy support at 12 months | 3 months and 12 months
  Important Other Climate Questionnaire adapted for physical activity and to query about one's team. Items rated on a Likert scale response format ranging from 1 (Strongly Disagree) to 7 (Strongly Agree) with a not applicable option, with higher total scores indicating higher perceived autonomy support.
Change in social support for physical activity at 3 months | Baseline and 3 months
  Social Support for Healthy Behaviors Questionnaire (physical activity support scale) adapted to query about one's team. Items scored using response options on a 5-point scale which ranges from almost never/not applicable to almost always, with higher mean scores indicating more support.
Change in social support for physical activity at 12 months | 3 months and 12 months
  Social Support for Healthy Behaviors Questionnaire (physical activity support scale) adapted to query about one's team. Items scored using response options on a 5-point scale which ranges from almost never/not applicable to almost always, with higher mean scores indicating more support.

OTHER OUTCOMES:
Mediation analysis of social support on moderate-to-vigorous intensity aerobic physical activity | 3 months and 12 months
  A mediation analysis will be conducted to explore whether social support mediates increased (at 3 months) and sustained (at 12 months) moderate-to-vigorous intensity aerobic physical activity within the overall study sample. The Social Support for Healthy Behaviors Questionnaire (physical activity support scale) adapted to query about one's team will be used to measure social support at baseline, 3 months, and 12 months. Items are scored using response options on a 5-point scale which ranges from almost never/not applicable to almost always, with higher mean scores indicating more support. Minutes per week of moderate-to-vigorous intensity aerobic physical activity will be measured using an accelerometer at baseline, 3 months, and 12 months. These data will facilitate the construction of mediation models.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Monroe, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article(s) reporting primary outcomes and secondary outcomes will be shared after deidentification. The study protocol, informed consent form, and statistical analysis plan will also be available to be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be made available 12 months after the publication of the article(s) that reported the data.
Access Criteria: Data will be made available via a study account posted on the Open Science Framework (https://www.osf.io)
URL: https://www.osf.io